CLINICAL TRIAL: NCT00217282
Title: Phase II Trial OF Oxaliplatin and Gemcitabine With Bevacizumab in Advanced Non-Small Cell Lung Cancer
Brief Title: Study of Oxaliplatin and Gemcitabine With or Without Bevacizumab to Treat Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Collaborators: Sanofi-Synthelabo (Industry); Genentech, Inc. (Industry)
Responsible Party: Rogerio Lilenbaum, Mount Sinai Medical Centent
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUN08
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Oxaliplatin; Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oxaliplatin, gemcitabine, bevacizumab — Gemcitabine 1000mg/m2 IV over 30 minutes, on days 1 and 8 followed by Oxaliplatin 130mg/m2 IV over 2 hours on day 1 followed by Bevacizumab 15 mg/kg IV over 90* minutes, on day 1 Cycles q 3 weeks x 4 cycles One cycle equals 3 weeks. Patients will be re-evaluated every 2 cycles. If CR, PR or SD, patients will continue treatment up to four cycles or until progression or unacceptable toxicity.
  Patients achieving CR, PR, or SD after 4 cycles will continue Bevacizumab maintenance:
  Bevacizumab 15 mg/kg IV q 3 weeks until relapse/progression

SUMMARY:
The combination of oxaliplatin and gemcitabine has proven activity in advanced non-small cell lung cancer (NSCLC). Due to its favorable toxicity profile, this combination is optimal for adding new agents. Bevacizumab is an anti-VEGF monoclonal antibody that has also shown favorable results in advanced NSCLC. This study will add bevacizumab to oxaliplatin and gemcitabine as first line treatment in patients with Stage IIIB and IV NSCLC.

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

Primary:

To determine the overall time to progression of the combination regimen of Gemcitabine, Oxaliplatin and Bevacizumab as first-line treatment in patients with Stage IIIB and IV non-small cell lung cancer.

Secondary

* To determine the overall response rate
* To determine the overall survival.
* To determine the toxicity of Gemcitabine, Oxaliplatin given in combination with Bevacizumab

ELIGIBILITY CRITERIA

1. Patients must have histologically or cytologically confirmed non-small cell lung cancer EXCEPT squamous cell carcinoma. Mixed tumors will be categorized by the predominant cell type unless small cell elements are present in which case the patient is ineligible. Cytologic or histologic elements can be established on metastatic tumor aspirates or biopsy.
2. Patients must have advanced NSCLC (Stage IIIB with malignant pleural effusion or Stage IV or recurrent disease).
3. Patients must have measurable disease (as defined in Section 13.0).
4. ECOG performance status 0 or 1.
5. Patients must not have known CNS metastases. Brain imaging is required within 4 weeks prior to study entry.
6. No prior systemic treatment for advanced NSCLC is permitted. Prior treatment for early-stage disease (adjuvant) or for locally-advanced Stage III disease is allowed if completed at least 12 months prior to registration.
7. Required laboratory values (obtained 2 weeks prior to registration):

   7.1 ANC > 1500/mm³. 7.2 Platelets > 100,000/mm³. 7.3 Total Bilirubin < 1.5 mg/dl. 7.4 Transaminases < 5 x ULN.
8. Patients must have adequate renal function as determined by the following tests within 2 weeks prior to registration.

   8.1 Serum creatinine less than or equal to 1.5 x upper limit of normal (ULN), AND Urinalysis < 1+ protein*

   * Patients discovered to have >1+ proteinuria at baseline must undergo a 24-hour urine collection. This must be an adequate collection and must demonstrate <1g of protein/24 hr to allow participation in the study.
9. Patients must be 18 years or older.
10. Pregnant and lactating women are excluded from the study because the agents used in this study may be teratogenic to a fetus and there is no information on the excretion of the agents or their metabolites into breast milk. A negative urine or serum pregnancy test required for women of childbearing potential.
11. Women of childbearing potential and sexually active males must agree to use an accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the study.
12. Patients treated with radiation therapy must have adverse events from therapy resolved to grade 2 or less following completion of treatment.
13. Patients must not have ongoing or active infection, symptomatic congestive heart failure, cerebrovascular accident within 12 months, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
14. Patients must have no deep vein thrombosis or pulmonary embolus within one year of registration and no ongoing need for full-dose oral or parenteral anticoagulation. Low dose coumadin (1mg) for maintenance of catheter patency or daily prophylactic aspirin is allowed.
15. Patients with history of hypertension must be well-controlled (defined as a blood pressure of >160 mmHg systolic and/or > 110 mmHg diastolic) on a stable regimen of anti-hypertensive therapy.
16. Patients must not have serious non-healing wound ulcer, or bone fracture, or major surgical procedure within 3 weeks prior to starting treatment.
17. Patients with a history of gross hemoptysis (defined as bright red blood of a ½ teaspoon or more) will be excluded from this trial
18. No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for five years

TREATMENT PLAN Gemcitabine 1000mg/m2 IV over 30 minutes, on days 1 and 8 followed by Oxaliplatin 130mg/m2 IV over 2 hours on day 1 followed by Bevacizumab 15 mg/kg IV over 90* minutes, on day 1 Cycles q 3 weeks x 4 cycles One cycle equals 3 weeks. Patients will be re-evaluated every 2 cycles. If CR, PR or SD, patients will continue treatment up to four cycles or until progression or unacceptable toxicity.

Patients achieving CR, PR, or SD after 4 cycles will continue Bevacizumab maintenance:

Bevacizumab 15 mg/kg IV q 3 weeks until relapse/progression

ELIGIBILITY:
Inclusion Criteria:

* Confirmed non-small cell lung cancer, EXCEPT squamous cell cancer
* Stage IIIB or IV disease
* ECOG PS 0-1
* No prior treatment
* No brain metastases
* Must have measurable disease

Exclusion Criteria:

* Deep vein thromboses or pulmonary embolus within 1 year
* History of gross hemoptysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To determine the overall time to progression of the combination regimen of Gemcitabine, Oxaliplatin and Bevacizumab as first-line treatment in patients with Stage IIIB and IV non-small cell lung cancer. | Prospective

SECONDARY OUTCOMES:
• To determine the overall response rate • To determine the overall survival. • To determine the toxicity of Gemcitabine, Oxaliplatin given in combination with Bevacizumab | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Lilenbaum, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, Miami Beach, Florida, United States